CLINICAL TRIAL: NCT04754230
Title: Effect of Tranexamic Acid on Postoperative Bleeding Following Sinus and Nasal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Zara M. Patel, Associated Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB-59164
Record Dates: First submitted 2021-02-10; First posted 2021-02-15 (Actual); Results first posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Chronic Sinusitis; Nasal Obstruction; Turbinate; Hypertrophy Mucous Membrane; Deviated Nasal Septum - Congenital; Deviated Nasal Septum Acquired
MeSH Terms: conditions — Nasal Obstruction | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1,000mg IV Tranexamic acid (Experimental): Participants in this arm will be given a 1,000mg dose of intravenous tranexamic acid via saline infusion 15 minutes prior to the completion of surgery. They will keep a bleeding diary with daily entries each day until their first routine scheduled postoperative follow-up clinic visit one week after surgery.
  Interventions: Drug: Tranexamic Acid 1,000 Mg/10 mL (100 Mg/mL) INTRAVEN VIAL (ML)
- Normal saline (No Intervention): Participants in this arm will not be given any extra intervention over their routine anesthetic care. They will continue to receive their normal saline infusion during surgery. They will keep a bleeding diary with daily entries each day until their first routine scheduled postoperative follow-up clinic visit one week after surgery.

INTERVENTIONS:
Drug: Tranexamic Acid 1,000 Mg/10 mL (100 Mg/mL) INTRAVEN VIAL (ML) — Medication administered 15 minutes prior to end of surgery.
  Arms: 1,000mg IV Tranexamic acid

SUMMARY:
The purpose of the research is to assess the effectiveness of a dose of intravenous tranexamic acid (TXA) given intraoperatively to reduce postoperative bleeding after endoscopic sinus or nasal surgery (e.g. septoplasty, endoscopic sinus surgery, turbinate surgery). This medication has been shown to decrease blood loss during this type of surgery, but the implications for bleeding following surgery are unclear. Any impact on postoperative bleeding will be assessed over the first 7 days following surgery leading up to the first scheduled postoperative clinic visit. Patients will keep a standardized daily diary of their bleeding experience by indicating on a 0-10 visual analog scale (VAS) their impression of their bleeding.

The primary outcome is the patient-reported visual analog scale (VAS) bleeding score on each day after surgery. The secondary outcomes include the the frequency with which the otolaryngology resident service is requested to evaluate patients in the recovery unit for postoperative bleeding concerns and the frequency of interventions such as application of hemostatic materials, packing, cautery, and/or return to the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo elective sinus or nasal surgery (e.g. septoplasty, inferior turbinate reduction, endoscopic sinus surgery)
* Age 18 or greater
* English-speaking
* Able to provide consent

Exclusion Criteria:

* Minors (age<18)
* Pregnant or may become pregnant by time of surgery
* Prisoners
* Non-English speaking
* Foreign citizens
* Unable to provide consent
* Known pro-thrombotic coagulation disorders
* Active intranasal drug use (e.g. cocaine)
* Surgery is for a sinonasal tumor or other sinus pathology not described in inclusion criteria
* Enrollment is in conflict with existing study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zara M. Patel, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

REFERENCES:
- [Background] Pundir V, Pundir J, Georgalas C, Fokkens WJ. Role of tranexamic acid in endoscopic sinus surgery - a systematic review and meta-analysis. Rhinology. 2013 Dec;51(4):291-7. doi: 10.4193/Rhino13.042. PMID 24260760
- [Background] Ping WD, Zhao QM, Sun HF, Lu HS, Li F. Role of tranexamic acid in nasal surgery: A systemic review and meta-analysis of randomized control trial. Medicine (Baltimore). 2019 Apr;98(16):e15202. doi: 10.1097/MD.0000000000015202. PMID 31008946
- [Background] Alimian M, Mohseni M. The effect of intravenous tranexamic acid on blood loss and surgical field quality during endoscopic sinus surgery: a placebo-controlled clinical trial. J Clin Anesth. 2011 Dec;23(8):611-5. doi: 10.1016/j.jclinane.2011.03.004. PMID 22137511
- [Background] Kim DH, Kim S, Kang H, Jin HJ, Hwang SH. Efficacy of tranexamic acid on operative bleeding in endoscopic sinus surgery: A meta-analysis and systematic review. Laryngoscope. 2019 Apr;129(4):800-807. doi: 10.1002/lary.27766. Epub 2018 Dec 28. PMID 30593688
- [Background] El-Ozairy HSE, Mady OM, Tawfik GM, Elhennawy AM, Teaima AA, Ebied A, Huy NT. Outcomes of combined use of topical and intravenous tranexamic acid on surgical field quality during functional endoscopic sinus surgery: Randomized controlled trial. Head Neck. 2021 May;43(5):1389-1397. doi: 10.1002/hed.26610. Epub 2021 Jan 31. PMID 33522019
- [Result] Khanwalkar A, Chan E, Roozdar P, Kim D, Ma Y, Hwang PH, Nayak JV, Patel ZM. Tranexamic acid does not significantly lower postoperative bleeding after endoscopic sinus and nasal surgery. Int Forum Allergy Rhinol. 2023 Sep;13(9):1584-1591. doi: 10.1002/alr.23127. Epub 2023 Feb 6. PMID 36608352

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline: Participants continue to receive their normal saline infusion during surgery.
- 1,000mg IV Tranexamic Acid: 1,000mg dose of intravenous tranexamic acid via saline infusion 15 minutes prior to the completion of surgery.
Period: Overall Study
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (16.2) | 41.5 (18.6) | 48.4 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 11 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bleeding VAS - POD1
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 1. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 1 (assessed within first 24 hours following surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 5.03 (2.14) | 4.82 (2.18)
Statistical Analysis 1: Comparison: Normal Saline vs 1,000mg IV Tranexamic Acid; Comparison of bleeding at day 1; Test type: Other; p = 0.8, two sided Z-test; This estimate uses two sided Z-test while assuming type I error=0.05

2. Primary Outcome: Bleeding VAS - POD2
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 2. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 4.47 (2.61) | 3.89 (2.01)

3. Primary Outcome: Bleeding VAS - POD3
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 3. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 2.93 (2.44) | 2.29 (1.21)

4. Primary Outcome: Bleeding VAS - POD4
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 4. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 2.12 (2.04) | 1.44 (1.23)

5. Primary Outcome: Bleeding VAS - POD5
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 5. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 1.32 (1.63) | 1.15 (0.94)

6. Primary Outcome: Bleeding VAS - POD6
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 6. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 1.36 (1.30) | 0.76 (0.83)

7. Primary Outcome: Bleeding VAS - POD7
Description: Patient-reported Visual Analog Scale - Bleeding Score Day 7. Score range: 0 (no bleeding) to 10 (uncontrolled bleeding).
Time Frame: Postoperative Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale | 0.97 (1.09) | 0.72 (0.89)

8. Secondary Outcome: Frequency of Participant Follow-up
Description: Number of patients in each arm requiring evaluation by the resident service for bleeding concerns expressed by the recovery nurse (in PACU), had any follow-up visit or phone call outside of regularly scheduled follow-up
Time Frame: Day of surgery through 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
Participants
  PACU | 0 | 0
  Follow-up visit | 0 | 1
  Follow-up phone call | 2 | 2

9. Primary Outcome: Guaze Saturation VAS Though POD7
Description: Patient-reported Visual Analog Scale - Guaze Saturation Score through Postoperative Day 7. Score range: 0 (not at all) to 10 (dripping blood).
Time Frame: Postoperative Day 2 through Postoperative Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
Number analyzed (Participants) | 19 | 21
score on a scale
  Postoperative day 2 | 5.16 (2.89) | 4.56 (2.50)
  Postoperative day 3 | 3.03 (3.05) | 2.09 (1.81)
  Postoperative day 4 | 1.74 (2.10) | 0.76 (1.34)
  Postoperative day 5 | 1.11 (1.56) | 0.40 (0.86)
  Postoperative day 6 | 0.99 (1.45) | 0.29 (1.81)
  Postoperative day 7 | 0.80 (1.05) | 0.28 (0.57)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Normal Saline | 1,000mg IV Tranexamic Acid
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT04754230/Prot_SAP_000.pdf